CLINICAL TRIAL: NCT04814095
Title: PRecision Oncology Evidence Development in Cancer Treatment - Clinical: PREDiCTc
Acronym: PREDiCTc
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PREDiCTc
Record Dates: First submitted 2021-03-01; First posted 2021-03-24 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Cancer
Keywords: targeted therapy; health technology assessment; real world evidence; quality of life
MeSH Terms: conditions — Neoplasms | interventions — Postmortem Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Targeted therapy (Experimental)
  Interventions: Behavioral: QOL; Diagnostic Test: CT imaging

INTERVENTIONS:
Behavioral: QOL — QOL assessments using the ESAS, CPC, EQ5D every 4-8 weeks +/- 2 weeks
Diagnostic Test: CT imaging — CT radiographic imaging every 12 weeks +/- 2 weeks

SUMMARY:
This pilot clinical trial aims to assess the real world quality of life and survival of patients treated with targeted therapy that has preliminary evidence of efficacy in subjects with advanced rare cancers or cancer harbouring rare molecular aberrations. The treatment has been granted conditional or full approved by Health Canada (HC) as effective and safe. Due to the rarity of the cancer or molecular aberration the uncertainty level of the health technology assessment (HTA) by the pan Canadian Oncology Review (pCODR) was too high for consideration of funding or it was not submitted for consideration. Consequently, the goal of this study is to generate real world evidence to support HTA decision making throughout the life cycle of the product.

DETAILED DESCRIPTION:
In Canada, adoption of new systemic therapies for cancer treatment is a multi-step process. After completion of clinical trials, pharmaceutical companies submit a request for a new drug approval to Health Canada. Therapies undergo rigorous review at Health Canada to confirm safety and efficacy before a Notice of Compliance (NOC) or NOC conditional (NOC/c) is issued that allows sale of the new medication in Canada. An additional layer of evaluation, a health technology assessment (HTA), is undertaken through the pan Canadian Oncology Drug Review (pCODR). A positive recommendation from pCODR is required for national price negotiations through the pan Canadian Pharmaceutical Alliance (pCPA). Once this step is completed, provincial pharmacies establish local contracts to permit local implementation of the new therapy.

As our understanding of pathogenesis evolves and next generation sequencing becomes more affordable, rare molecular entities amenable to treatment with targeted or selected therapies, like immunotherapy, are being increasingly identified. These molecular aberrations can occur with frequencies of 1-2% making it unfeasible to conduct large randomized trials to establish benefit. Determination of the added value of these new therapies in terms of outcomes and quality of life is challenging in the absence of comparators in trials resulting in increased uncertainty in terms of outcomes, quality of life (QOL) and cost-effectiveness. To address the uncertainty, pharmaceutical companies and the pCODR economic guidance panel create economic models with sensitivity analyses to try to estimate the cost-effectiveness of therapy. These models however, are dependent on the nature and quality of available data.

This study proposes to use real world data to generate evidence to assist in evaluate new therapies in rare molecular entities. The key components include regular interval radiographic imaging and collection of patient reported outcomes using standardized QOL questionnaires. The aim is to provide high quality real world evidence for assessment and economic modelling to reduce uncertainty and facilitate HTA decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Subject age greater than or equal to 18 years at the time of signature of informed consent.
* Subjects with an incurable malignancy who have been identified to have a rare cancer or rare molecular aberration who is currently receiving Health Canada approved targeted therapy that is not nationally funded
* ECOG 0-2
* Life expectancy of at least 12 weeks
* Adequate hematologic and end organ function for drug treatment per the clinician's assessment
* Asymptomatic or treated brain metastases permitted
* Ability to give informed consent for the study procedures defined in this protocol.

Exclusion Criteria:

* Treatment with any approved or investigational agent or participation in another clinical trial with therapeutic intent within 14 days prior to enrollment.
* Inability to complete quality of life questionnaires
* Subjects who are felt by the treating clinician to be unfit to proceed with this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival from initiation of targeted therapy | Baseline until death up to 5 years

SECONDARY OUTCOMES:
Response rate as defined by RECIST 1.1 | Baseline until progression up to 5 years
Response rate as defined by physician assessed response | Baseline until progression up to 5 years
Progression free survival (PFS) from initiation of targeted therapy | Baseline until progression up to 5 years
Quality of life (QoL) assessments using the EQ-5D every 8 weeks from initiation of targeted therapy | Baseline until death up to 5 years
Quality adjusted survival from initiation of targeted therapy | Baseline until death up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Ho, MD, Principal Investigator — BC Cancer
Locations (1):
- BC Cancer, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No